CLINICAL TRIAL: NCT03852771
Title: CompRESsion Therapy for Restless Leg Syndrome: An Evaluation of Cirvo™ for the Treatment of Restless Leg Syndrome
Brief Title: REST Study (CompRESsion Therapy for RLS)
Acronym: REST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company closure
Sponsor: Radial Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-00383
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-03

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): All participants will receive the intervention
  Interventions: Device: Cirvo(TM) therapy

INTERVENTIONS:
Device: Cirvo(TM) therapy — The Cirvo(TM) (also referred to as the Radial Medical Compression System) is a mobile wearable medical device that applies graded intermittent mechanical sequential compression to the lower leg.

SUMMARY:
This study in patients with restless leg syndrome (RLS) will evaluate the use of Cirvo™ therapy for the treatment of this disorder when applied to both legs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over the age of 18.
2. Diagnosis of Restless Leg Syndrome (RLS) per the Hopkins-Hening Diagnostic Questionnaire
3. International RLS Study Group (IRLSS) Score ≥15.
4. RLS symptoms occurring on at least 5 nights each week, with symptoms stable for at least 3 months.

Exclusion Criteria:

1. Known or suspected deep vein thrombosis.
2. Pregnancy
3. Prior use with home intermittent pneumatic compression (IPC) device
4. Currently using any other device to treat RLS
5. Active skin infections in the affected leg
6. Vein ligation or skin graft of the leg within past 12 months
7. Mental or physical limitations that would prevent the subject from reliably completing study questionnaires.
8. Physical impairments that would prevent the use of the CirvoTM device.
9. Use of any medications typically used to treat RLS, where dose has not been stable for at least 2 months.
10. If previously on medication to treat RLS, patient must have been weened under medical supervision and off medication for at least 14 days at time of enrollment
11. History of pulmonary vascular disease (PVD)
12. History of pulmonary edema
13. History of decompensated congestive heart failure (CHF)
14. Open surgery or major trauma to the legs within the last six months
15. History of lower limb malignancy, primary or secondary
16. Acute symptomatic lower extremity thrombophlebitis
17. Any chronic back pain or lower extremity pain
18. Other sleep problems that are felt to be currently affecting the quality of sleep
19. Calf geometry on which Cirvo™ device does not appropriately fit
20. Known sensitivity to any of the materials used in the Cirvo™ device
21. Currently participating or plans to participate in in any other investigational clinical evaluation during the 56 day study period that may, in the opinion of the investigator, affect RLS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in disease severity between the Baseline study visit and the 56-day visit, as assessed by the International Restless Leg Syndrome Study Group Severity Scale (IRLSS). | 56 days
  Assessment of change in IRLSS scores from Baseline study visit to 56 days.

SECONDARY OUTCOMES:
Change in disease severity between the Baseline study visit and the 56-day visit, as assessed by the Clinical Global Impression (CGI-I) rating scale. | 56 days
  Change in disease severity as assessed by CGI-I scale
Change in sleep quality between the Baseline study visit and the 56-day visit, as assessed by the Medical Outcomes Study (MOS) sleep scale. | 56 days
  Change in sleep quality as assessed by MOS sleep scale from Baseline to 56 days
Change in disease severity between the Baseline study visit and after the last usage of the each parameter set trialed in Period 1 (nominally days 7, 14, 21, and 28), as assessed by the IRLSS. | 28 days
  Assessment of IRLSS score after each week of programmed therapy for first 4 weeks of therapy.

OTHER OUTCOMES:
Therapy related adverse events | 56days
  Assessment of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- California Center for Sleep Disorders, Alameda, California, United States

IPD SHARING:
Plan to Share IPD: No